CLINICAL TRIAL: NCT00340860
Title: The Norwegian Mother and Child Study - Environmental Specimen Collection
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902206; 02-E-N206
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Environmental Determinants; Pregnancy
Keywords: Disease Activity; Pregnancy; Exposure; Norway Mother and Child Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Norweigian Population-Based Pregnancy Cohort: Norwegian-speaking pregnant women, their children born post enrollment, and enrolled children's fathers

SUMMARY:
The Norway Mother and Child study is a collaborative venture among health researchers in Norway funded by the Norwegian government. The study is being coordinated by the National Institute of Public Health (aka Folkehelsa) in Oslo and the Medical Birth Registry (MBR) in Bergen. NIEHS has the unique opportunity to participate through the collection of additional tubes of blood during the blood sample collection; these two tubes of blood and a urine sample will allow NIEHS and collaborators to explore environmental determinants for disease among women and their children. These additional samples will remain in the Biobank in Oslo, Norway, with other samples from cohort members and will be used under collaboration with Norwegian investigators.

To achieve better health for mothers and children in the future, the Norway Mother and Child study is designed to test specific hypotheses about the causes of a number of serious diseases by recruiting 110,000 pregnant women to a cohort study. As part of the primary aim of the study, women will be asked to provide a blood sample at 17 weeks gestation, at birth, and 4 days after birth. The NIEHS samples will be collected at the blood draw at 17 weeks gestation. Likely causal factors will be linked to information obtained from questionnaires, blood samples, and medical registers.

The Norway Mother and Child study has multiple endpoints. Primarily those associated with adverse pregnancy outcomes will be studied, but also diseases affecting mother, father or child. Endpoints will be taken from questionnaires and medical registers. The study will be carried out nationally and any research groups with relevant questions will be able to participate. The Norway Mother and Child study has been approved by the Norwegian Parliament as well as their Data Inspectorate to ensure that the study and all protocols conform to Norwegian ethical standards as well as appropriate research ethical criteria. Further, the project has been evaluated by the Regional Ethics Committee for Medical Research which has approved all modifications to the project.

Other researchers, nationally and internationally, will have access to the cohort on request and following approval from the project's executive group. NIEHS has the opportunity to add additional biological specimens for blood and urine to the base cohort. Two additional tubes of blood (total volume 9 ml) and a urine sample will be collected as part of the routine prenatal ultrasound visit and blood sample collection included in the overall study protocol. As part of a reliability sub-study, blood and urine samples will also be collected an additional two times, at weeks 23 and 29 of gestation. These samples are designed to allow investigators to explore environmental contributors to the health of women and their children. Low level exposure to environmental contaminants occurs in all industrialized countries, though the level of exposure may differ as the result of diet, cooking practices and pollution sources. However, the ability to explore the role of environmental exposure on health is often more limited by good population-based information on health and disease then by exposure level. Thus, by creating a biological specimen repository in a country with excellent disease registries, it will allow NIEHS to explore risk factors for disease relevant to US populations. All samples will be stored in Norway and will be used in collaboration with Norwegian and other investigators. NIEHS investigators will not have access to identifying information. NIEHS samples will not be used for genetic analyses.

...

DETAILED DESCRIPTION:
The Norway Mother and Child study is a collaborative venture among health researchers in Norway funded by the Norwegian government. The study is being coordinated by the National Institute of Public Health (aka Folkehelsa) in Oslo and the Medical Birth Registry (MBR) in Bergen. NIEHS has the unique opportunity to participate through the collection of additional tubes of blood during the blood sample collection; these two tubes of blood and a urine sample will allow NIEHS and collaborators to explore environmental determinants for disease among women and their children. These additional samples will remain in the Biobank in Oslo, Norway, with other samples from cohort members and will be used under collaboration with Norwegian investigators.

To achieve better health for mothers and children in the future, the Norway Mother and Child study is designed to test specific hypotheses about the causes of a number of serious diseases by recruiting 110,000 pregnant women to a cohort study. As part of the primary aim of the study, women will be asked to provide a blood sample at 17 weeks gestation, at birth, and 4 days after birth. The NIEHS samples will be collected at the blood draw at 17 weeks gestation. Likely causal factors will be linked to information obtained from questionnaires, blood samples, and medical registers.

The Norway Mother and Child study has multiple endpoints. Primarily those associated with adverse pregnancy outcomes will be studied, but also diseases affecting mother, father or child. Endpoints will be taken from questionnaires and medical registers. The study will be carried out nationally and any research groups with relevant questions will be able to participate. The Norway Mother and Child study has been approved by the Norwegian Parliament as well as their Data Inspectorate to ensure that the study and all protocols conform to Norwegian ethical standards as well as appropriate research ethical criteria. Further, the project has been evaluated by the Regional Ethics Committee for Medical Research which has approved all modifications to the project.

Other researchers, nationally and internationally, will have access to the cohort on request and following approval from the project's executive group. NIEHS has the opportunity to add additional biological specimens for blood and urine to the base cohort. Two additional tubes of blood (total volume 9 ml) and a urine sample will be collected as part of the routine prenatal ultrasound visit and blood sample collection included in the overall study protocol. As part of a reliability sub-study, blood and urine samples will also be collected an additional two times, at weeks 23 and 29 of gestation. These samples are designed to allow investigators to explore environmental contributors to the health of women and their children. Low level exposure to environmental contaminants occurs in all industrialized countries, though the level of exposure may differ as the result of diet, cooking practices and pollution sources. However, the ability to explore the role of environmental exposure on health is often more limited by good population-based information on health and disease then by exposure level. Thus, by creating a biological specimen repository in a country with excellent disease registries, it will allow NIEHS to explore risk factors for disease relevant to US populations. All samples will be stored in Norway and will be used in collaboration with Norwegian and other investigators. NIEHS investigators will not have access to identifying information. NIEHS samples will not be used for genetic analyses.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study sample will be all pregnant women scheduled for routine ultrasound at 16-18 weeks gestation.

EXCLUSION CRITERIA:

Women who do not speak Norwegian are excluded because they cannot complete the questionnaires.

RELIABILITY SUB-STUDY ELIGIBILITY CRITERIA:

Subjects must be enrolled in the Norway Mother and Child Study at one of four participating hospitals and have successfully completed a blood draw and urine collection in the 17th week of gestation.

SEVEN-YEAR FOLLOW-UP PILOT STUDY ELIGIBILITY CRITERIA:

Mothers and children must be enrolled in the Norway Mother and Child Study and the child must turn seven years of age during pilot enrollment in 2008 and 2009.

Ages: 15 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Norwegian pregnant women are prospectively followed beginning with the 17th week of pregnancy. Their children born after enrollment are prospectively followed into adulthood. Enrolled children's fathers are prospectively followed as well.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 81093 (Actual)
Dates: Start 2001-10-01 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
NIEHS samples will be used to assess the role of environmental exposures on health | 17, 23, and 29 weeks gestation
  Adverse pregnancy outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gitanjali Taneja, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- Norwegian Institute of Public Health and Birth Registry, Bergen, Norway